CLINICAL TRIAL: NCT03521063
Title: Efficacy of Adding Budesonide to Poractant Alfa to Prevent Bronchopulmonary Dysplasia in Preterm Infants With Respiratory Distress Syndrome.
Brief Title: Efficacy of Adding Budesonide to Poractant Alfa to Prevent Bronchopulmonary Dysplasia.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Collaborators: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Raúl Héctor Roque Sánchez, MD, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 86-17
Record Dates: First submitted 2018-04-28; First posted 2018-05-11 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Bronchopulmonary Dysplasia; Infant,Premature; Respiratory Distress Syndrome
Keywords: bronchopulmonary dysplasia; respiratory distress syndrome; budesonide; poractant alfa
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Respiratory Distress Syndrome | interventions — Budesonide; poractant alfa; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Poractant alfa/budesonide (Experimental): A mixture of poractant (200mg/kg) and budesonide (0.25 mg/kg) will be instilled intratracheal
  Interventions: Drug: Budesonide; Drug: Poractant Alfa
- Poractant alfa/saline (Active Comparator): A mixture of poractant (200mg/kg) and saline (1 ml/kg) will be instilled intratracheal
  Interventions: Drug: Poractant Alfa; Drug: Saline

INTERVENTIONS:
Drug: Budesonide — Drug: Budesonide inhalation suspension
  Other Names: Pulmicort
  Arms: Poractant alfa/budesonide
Drug: Poractant Alfa — Drug: Poractant alfa intratracheal suspension
  Other Names: Curosurf
Drug: Saline — Sodium chloride injection 0.9%
  Other Names: Normal saline
  Arms: Poractant alfa/saline

SUMMARY:
This study evaluates the addition of budesonide to poractant alfa to prevent bronchopulmonary dysplasia in preterm infants with respiratory distress syndrome. Half of the participants will receive budesonide and poractant alfa in combination, and the other half will receive poractant alfa with saline.

DETAILED DESCRIPTION:
A randomized double bind controlled trial, designed to evaluate the addition of budesonide to poractant alfa to prevent bronchopulmonary dysplasia (BPD) in preterm infants with respiratory distress syndrome (RDS).

The usual treatment of RDS includes ventilatory support and exogenous surfactant, however, a cronic lung disease known as BPD, is a complication found in many of these patients.

BPD is a complex disease occurring in preterm infants recovering from RDS and inflammation plays a key role in its physiopathology.

Animal derived surfactants have demonstrated to decrease the incidence of BPD, and porcine surfactant (poractant alfa) has and increased effect compared with bovine surfactant (beractant).

Budesonide is an inhaled anti-inflammatory steroid that has shown to reduce BPD when combined with beractant by decreasing lung inflammation, without secondary systemic effects, when combined with poractant alfa it could enhance even more this anti-inflammatory effect.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <1500g
* Gestational age ≥ 26 weeks
* Respiratory distress syndrome that requires exogenous surfactant at birth or in the first 12 hours of life.

Exclusion Criteria:

* Major congenital anomalies.
* Perinatal asphyxia
* Respiratory depression secondary to general anesthesia.

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia or death | Oxygen requirement at 36 weeks post menstrual age in patients <32 weeks. Oxygen requirement between 29 to 55 days of age in patients >32 weeks
  Diagnosis of bronchopulmonary dysplasia according to NICHD criteria

CONTACTS AND LOCATIONS:
Overall Officials: RAUL H ROQUE SANCHEZ, MD, Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Halliday HL; European Association of Perinatal Medicine. European consensus guidelines on the management of neonatal respiratory distress syndrome in preterm infants--2013 update. Neonatology. 2013;103(4):353-68. doi: 10.1159/000349928. Epub 2013 May 31. PMID 23736015
- [Background] Singh N, Halliday HL, Stevens TP, Suresh G, Soll R, Rojas-Reyes MX. Comparison of animal-derived surfactants for the prevention and treatment of respiratory distress syndrome in preterm infants. Cochrane Database Syst Rev. 2015 Dec 21;2015(12):CD010249. doi: 10.1002/14651858.CD010249.pub2. PMID 26690260
- [Background] Yeh TF, Chen CM, Wu SY, Husan Z, Li TC, Hsieh WS, Tsai CH, Lin HC. Intratracheal Administration of Budesonide/Surfactant to Prevent Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2016 Jan 1;193(1):86-95. doi: 10.1164/rccm.201505-0861OC. PMID 26351971
- [Background] Venkataraman R, Kamaluddeen M, Hasan SU, Robertson HL, Lodha A. Intratracheal Administration of Budesonide-Surfactant in Prevention of Bronchopulmonary Dysplasia in Very Low Birth Weight Infants: A Systematic Review and Meta-Analysis. Pediatr Pulmonol. 2017 Jul;52(7):968-975. doi: 10.1002/ppul.23680. Epub 2017 Feb 6. PMID 28165675